CLINICAL TRIAL: NCT07237906
Title: Neutropenia in Patients Treated With TNF-α Inhibitors: Frequency and Clinical Implications From a Retrospective Cohort
Brief Title: Neutropenia With TNF-α Inhibitors
Status: Completed | Type: Observational
Sponsor: Burak Ugur Cetin (Other)
Responsible Party: Sponsor-Investigator, Burak Ugur Cetin, Medical Doctor, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Other Study IDs: IstanbulUC-BCetin-02
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Neutropenia; TNF-alpha Inhibitors
Keywords: Adverse drug event; Arthritis; Neutropenia; Tumor necrosis factor-alpha inhibitors
MeSH Terms: conditions — Neutropenia; Drug-Related Side Effects and Adverse Reactions; Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group: Patients receiving TNF-α inhibitor therapy for inflammatory arthritis

SUMMARY:
Tumor necrosis factor-alpha (TNF-α) inhibitors, including infliximab, etanercept, adalimumab, certolizumab, and golimumab, have become cornerstone therapies in the management of rheumatologic disorders. Although their efficacy and tolerability are well established, accumulating evidence indicates that these agents may also induce hematologic adverse events. The most frequently documented hematologic complication of TNF-α inhibitor therapy is neutropenia. Previous studies have reported neutropenia in approximately 10-19% of patients receiving TNF-α inhibitors.

Neutropenia is defined as a decrease in circulating neutrophils to an absolute neutrophil count (ANC) below 1500 cells/μL. Clinically, neutropenia is stratified according to the ANC as mild (1000-1500/μL), moderate (500-1000/μL), or severe (<500/μL). While mild neutropenia is frequently asymptomatic, severe neutropenia is associated with a substantially elevated risk of serious and potentially life-threatening infections .

The pathophysiological mechanisms underlying drug-induced neutropenia remain incompletely understood; however, proposed explanations include immune-mediated peripheral destruction of granulocytes, bone marrow suppression or impaired maturation of granulocyte precursors. Autoimmune pathways may also contribute, as evidenced by recurrence of neutropenia following drug rechallenge.

Neutropenia associated with TNF-α inhibitor therapy is typically mild; however, its development warrants careful clinical attention. Certain clinical risk factors have been identified. Identified risk factors include a previous history of neutropenia, prior neutropenia under disease-modifying antirheumatic drugs (DMARDs) therapy, and lower baseline neutrophil counts, each of which may predispose patients to subsequent neutropenia. Notably, most cases emerge within the first three months after treatment initiation. Although discontinuation is rarely required and serious infections are uncommon, the possibility of hematologic complications underscores the importance of close monitoring and routine hematologic assessments throughout therapy. Despite the growing recognition of TNF-α inhibitor-induced neutropenia, current data regarding its rate, clinical course, and impact on treatment outcomes remain limited, particularly in real-world patient populations. The present study aimed to determine the frequency of neutropenia in this population and to evaluate its clinical characteristics and impact on treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of TNF-alpha inhibitor therapy at least once in our clinic between September 2023 and January 2025
* Age 18 years or older
* At least one complete blood count performed during the follow-up period
* Availability of complete clinical and laboratory data in the hospital's electronic medical records or patient files

Exclusion Criteria:

* History of other hematologic disorders that may contribute to the development of neutropenia (e.g., aplastic anemia, leukemia, myelodysplastic syndrome)
* Concurrent treatment with cytotoxic chemotherapy or immunosuppressive agents (e.g., azathioprine, cyclophosphamide)
* Insufficient follow-up duration or incomplete laboratory data that precluded adequate evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory arthritis who were treated with TNF-α inhibitor therapy at the Physical Medicine and Rehabilitation Department of Istanbul University-Cerrahpasa, a tertiary care center in Istanbul, Turkey, between September 2023 and January 2025.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of neutropenia | From initiation of TNF-α inhibitor therapy to 12 months of treatment
  Incidence of neutropenia in patients receiving TNF-α inhibitors

SECONDARY OUTCOMES:
Severity of neutropenia | From initiation of TNF-α inhibitor therapy to 12 months of treatment
  Clinically, neutropenia is stratified according to the ANC as mild (1000-1500/μL), moderate (500-1000/μL), or severe (<500/μL).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a retrospective, single-center study based on patient records. Due to privacy concerns and institutional regulations, individual participant data will not be shared.